CLINICAL TRIAL: NCT02839707
Title: A Randomized, Phase II/III Study of Pegylated Liposomal Doxorubicin and CTEP-Supplied Atezolizumab Versus Pegylated Liposomal Doxorubicin, CTEP-Supplied Bevacizumab and CTEP-Supplied Atezolizumab Versus Pegylated Liposomal Doxorubicin and CTEP-Supplied Bevacizumab in Platinum Resistant Ovarian Cancer
Brief Title: Pegylated Liposomal Doxorubicin Hydrochloride With Atezolizumab and/or Bevacizumab in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01081; NCI-2016-01081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY009; NRG-GY009 (Other: NRG Oncology); NRG-GY009 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-07-20; First posted 2016-07-21 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Fallopian Tube High Grade Serous Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Fallopian Tube Clear Cell Adenocarcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Fallopian Tube Undifferentiated Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian Undifferentiated Carcinoma; Recurrent Platinum-Resistant Fallopian Tube Carcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Clear Cell Adenocarcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal Undifferentiated Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (PLD, atezolizumab) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and atezolizumab IV over 30-60 minutes on days 1 and 15. (Closed to accrual as of February 09, 2021)
  Interventions: Drug: Atezolizumab; Procedure: Computed Tomography; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment
- Arm II (PLD, bevacizumab, atezolizumab) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1, bevacizumab IV over 30-90 minutes on days 1 and 15, and atezolizumab IV over 30-60 minutes on days 1 and 15. Patients also undergo CT on study.
  Interventions: Drug: Atezolizumab; Biological: Bevacizumab; Procedure: Computed Tomography; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment
- Arm III (PLD, bevacizumab) (Active Comparator): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and bevacizumab IV over 30-90 minutes on days 1 and 15. Patients also undergo CT on study.
  Interventions: Biological: Bevacizumab; Procedure: Computed Tomography; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm I (PLD, atezolizumab); Arm II (PLD, bevacizumab, atezolizumab)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm II (PLD, bevacizumab, atezolizumab); Arm III (PLD, bevacizumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II/III trial studies how well pegylated liposomal doxorubicin hydrochloride with atezolizumab and/or bevacizumab work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back (recurrent). Chemotherapy drugs, such as pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. It is not yet known which combination will work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the probability of a dose limiting toxicity (DLT) following cycle 1 of experimental regimens (pegylated liposomal doxorubicin hydrochloride [pegylated liposomal doxorubicin] [PLD] and atezolizumab and PLD/bevacizumab and atezolizumab). (Safety lead-in) II. Estimate and compare the hazard of first progression or death (progression free survival [PFS]) of each experimental regimen relative to the reference regimen, PLD and bevacizumab. (Phase II study) III. Estimate and compare the hazard of death and the hazard of first progression or death (PFS) of the experimental regimen relative to the reference regimen. (Phase III) (24-FEB-2021)

SECONDARY OBJECTIVES:

I. Estimate and compare the probabilities of response (objective response rate [ORR], either partial or complete response) defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria on each study regimen. (Phase II study) (24-FEB-2021) II. Estimate the frequency and severity of adverse events as classified and graded with Common Terminology Criteria for Adverse Events (CTCAE) in those patients who initiate their randomly assigned study treatment. (Phase II study) (03/19/2018) III. Estimate and compare ORR in each treatment group. (Phase III study) IV. Estimate the frequency and severity of adverse events in those patients who initiate their randomly assigned study treatment. (Phase III study) V. Estimate and compare mean patient reported outcome scores (PROs) as measured by National Comprehensive Cancer Network (NCCN)-Functional Assessment of Cancer Therapy (FACT) ovarian symptom index (NFOSI)-18 disease-related symptoms (DRS). (Phase III study) VI. Estimate and compare the treatment groups on the basis of the PROs: treatment side effects (TSE), function/well-being (FWB), fatigue (Functional Assessment of Chronic Illness Therapy [FACIT]-fatigue subscale) and abdominal discomfort (FACT/Gynecologic Oncology Group [GOG]-abdominal discomfort [AD] subscale). (Phase III study) (10/16/2017)

TRANSLATIONAL SCIENCE OBJECTIVES:

I. To determine whether biomarker levels in pre-treatment tissue, and pre- or on-treatment peripheral blood, and stool specimens are associated with ORR, PFS and/or overall survival (OS).

II. Estimate pre-treatment PD-L1 expression on tumor cells measured by quantitative immunohistochemistry (IHC), and determine whether it is associated with the duration of PFS or overall survival. (Integrated Biomarker) III. Analysis of T cell receptor (TCR) repertoires by deep sequencing of peripheral blood samples. (Exploratory Biomarkers [10/16/2017]) IV. Tumor "immunogenicity" as determined by the neo-antigen landscape and characterization of the tumor microenvironment using next-generation sequencing, including but not limited to whole exome sequencing and/or RNA sequencing. (Exploratory Biomarkers [10/16/2017]) V. Microbiome analysis via stool sampling. (Exploratory Biomarkers [10/16/2017]) VI. To determine whether changes in quantitative biomarker parameters after the first 6 and 12 weeks of therapy predict ORR, PFS and/or OS.

OUTLINE: Patients will be randomized to 1 of 3 arms.

ARM I: Patients receive pegylated liposomal doxorubicin hydrochloride intravenously (IV) over 60 minutes on day 1 and atezolizumab IV over 30-60 minutes on days 1 and 15. (Closed to accrual as of February 09, 2021)

ARM II: Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1, bevacizumab IV over 30-90 minutes on days 1 and 15, and atezolizumab IV over 30-60 minutes on days 1 and 15. Patients also undergo computed tomography (CT) on study.

ARM III: Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and bevacizumab IV over 30-90 minutes on days 1 and 15. Patients also undergo CT on study.

In all arms, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up
* Administration of study drugs (pegylated liposomal doxorubicin, bevacizumab, atezolizumab) may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. (06/29/2017)
* Submission of tumor tissue is required for all patients; investigators should check with their site pathology department regarding release of biospecimens before approaching patients about participation in the trial
* High grade ovarian cancer, including high grade serous; clear cell; endometrioid, grade 3; and others (adenocarcinoma, not otherwise specified [NOS]; mixed epithelial carcinoma; undifferentiated carcinoma); NOTE: low grade serous, mucinous and carcinosarcoma histologies are excluded due to their different underlying genomic features and/or clinical behavior; ovarian cancer = ovarian, fallopian tube or primary peritoneal cancer; required data element: submission of pathology report
* Recurrent, platinum resistant ovarian cancer (defined as progression within < 6 months from completion of platinum based therapy; the date should be calculated from the last administered dose of platinum therapy)
* 1-2 prior regimens (including primary therapy); hormonal therapies (e.g., tamoxifen, aromatase inhibitors) will not count toward the prior regimen limit; PARP inhibitors given in the maintenance setting post response to platinum-based therapy will not count as a separate regimen from the preceding platinum-based therapy. (30-OCT-2020)
* Measurable disease (defined by RECIST v1.1) or evaluable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease related in the setting of cancer antigen [CA] 125 >= 2 x upper limit of normal [ULN])
* Age >= 18
* Performance status 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to registration)
* Platelets >= 100,000/mcl (within 14 days prior to registration)
* Hemoglobin (Hgb) >= 8 g/dl (within 14 days prior to registration)
* Creatinine =< 1.5 x institutional upper limit of normal (ULN) (within 14 days prior to registration)
* Urine protein creatinine (UPC) ratio must be < 1.0 (within 14 days prior to registration); if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended (24-hour urine protein level must be < 1000 mg for patient enrollment); If UPC ratio cannot be calculated because the urine protein is below the lower limit of detection of the assay this will not exclude the patient (10/22/2018) (30-OCT-2020); UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* Total bilirubin =< 1.5 x ULN (patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled) (within 14 days prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement) (within 14 days prior to registration)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (or on stable dose of therapeutic anticoagulation, such as low-molecular-weight heparin, warfarin or rivaroxaban) (10/16/2017)
* Thyroid-stimulating hormone (TSH) within normal limits (Euthyroid patients on thyroid replacement therapy allowed provided TSH < ULN) (02/20/2019)
* The patient or legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients who have had systemic anticancer therapy (e.g., chemotherapy, targeted therapy including PARP inhibitors or bevacizumab) within 3 weeks prior to entering the study (30-OCT-2020)
* Patients who have had hormonal therapy (e.g., tamoxifen, aromatase inhibitor) within 1 week prior to entering the study
* Patients with prior treatment with anti-programmed cell death (PD)-1, anti- programmed cell death ligand (PD-L)1 or anti-cytotoxic T-lymphocyte-associated protein (CTLA)-4 therapeutic antibody or other similar agents (10/16/2017)
* Patients with prior treatment with bevacizumab (or any other anti vascular therapy, e.g., cediranib) for platinum resistant recurrence; (Note: prior bevacizumab in initial therapy and/or platinum sensitive recurrent setting is allowed) (10/16/2017)
* Patients with prior treatment with PLD
* Prior radiotherapy to the abdomen or pelvis
* Patients who have not recovered from adverse events to =< grade 1 (other than alopecia) due to agents administered more than 3 weeks earlier (10/16/2017); however, the following therapies are allowed:

  * Hormone replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to cycle 1, day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to cycle 1, day 1)
  * Palliative radiotherapy for bone metastases > 2 weeks prior to cycle 1, day 1
* Treatment with any other investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea or steroids as computed tomography [CT] scan contrast premedication) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia within the past 28 days; use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy within 28 days prior to cycle 1, day 1
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to cycle 1, day 1
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients requiring treatment with a receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis (02/20/2019)

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen, or type 2 diabetes mellitus are eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab (06/29/2017)

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial (08-JAN-2021)
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years, with the exception of those with a negligible risk of metastases or death, such as carcinoma in situ of the breast or cervix
* Severe, active co-morbidity defined as follows:

  * Current (within 28 days of cycle 1, day 1) signs and/or symptoms of bowel obstruction
  * Patients who require parental hydration and/or nutrition
  * Patients who require drainage gastrostomy tube
  * Evidence of bleeding diathesis or clinically significant coagulopathy
  * Serious, non-healing or dehiscing wound, active ulcer or untreated bone fracture
  * History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment
* Significant cardiovascular or cerebrovascular disease including:

  * Uncontrolled hypertension (systolic blood pressure [SBP] >= 150 and/or diastolic blood pressure [DBP] >= 90)
  * History of myocardial infarction within 6 months
  * Unstable angina
  * New York Heart Association functional classification II, III or IV
  * Baseline ejection fraction =< 50% as assessed by echocardiogram or multi-gated acquisition (MUGA)
  * Cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months
  * Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or peripheral arterial thrombosis) within 6 months
* History of abdominal/pelvic or tracheoesophageal fistula or gastrointestinal perforation and/or abdominal/pelvic abscess within 6 months prior to initiation of treatment (02/20/2019)
* Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin E O'Cearbhaill, Principal Investigator — NRG Oncology
Locations (922):
- United States (910):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Valley Medical Group - Wayne Multispecialty Practice, Wayne, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Medical Center Clinic-New Castle Office, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Gynecologic Oncology, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (12):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from June of 2017 to October of 2021.
Period: Phase I
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Started | 17 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 9 | 0 | 0
Not completed — Not eligible for analysis | 9 | 0 | 0
Period: Phase II
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Started | 80 | 80 | 80
Completed | 76 | 80 | 78
Not Completed | 4 | 0 | 2
Not completed — Not treated according to protocol | 4 | 0 | 2
Period: Phase III
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Started | 27 | 72 | 72
Completed | 27 | 72 | 68
Not Completed | 0 | 0 | 4
Not completed — Not treated according to protocol | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab) | Total
Number analyzed (Participants) | 124 | 160 | 160 | 444
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 62 [55 to 68] | 64 [56 to 70] | 63 [56 to 69] | 63 [56 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 160 | 160 | 444
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 8 | 29
  Not Hispanic or Latino | 113 | 147 | 149 | 409
  Unknown or Not Reported | 1 | 2 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 7 | 9 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 14 | 11 | 35
  White | 104 | 133 | 130 | 367
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 6 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLT) of Experimental Regimens
Description: Will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 (CTCAE version 5.0 will be used beginning April 1, 2018). DLT will be assessed.
Time Frame: Up to 28 days
Population: Patients enrolled into safety stage 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 17 | 8 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria and will include estimates of the hazard ratios and the corresponding confidence intervals for the experimental regimen relative to the reference regimen, as well as Kaplan-Meier estimates of the survivorship function for each treatment group. Progression is defined by a 20% increase in the sum of the longest diameter of target lesions and a 5 mm absolute increase from nadir, or an unequivocal increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From study enrollment to the investigator determined date of progression or death due to any cause, whichever occurs first, assessed up to 5 years
Population: Eligible patients enrolled in Phase I and II.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (PLD, Atezolizumab): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and atezolizumab IV over 30-60 minutes on days 1 and 15. (Closed to accrual as of February 09, 2021) Atezolizumab: Given IV Computed Tomography: Undergo CT Pegylated Liposomal Doxorubicin Hydrochloride: Given IV Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 88 | 88 | 88
months | 4.2 [3.4 to 5.6] | 7.6 [5.6 to 8.8] | 5.5 [3.9 to 7.3]

3. Primary Outcome: PFS (Phase III)
Description: Will be assessed by RECIST v1.1 criteria and will include estimates of the hazard ratios and the corresponding confidence intervals for the experimental regimen relative to the reference regimen, as well as Kaplan-Meier estimates of the survivorship function for each treatment group.
  Progression is defined by a 20% increase in the sum of the longest diameter of target lesions and a 5 mm absolute increase from nadir, or an unequivocal increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 2
Population: Eligible patients enrolled in Phase I, II and III.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 115 | 160 | 160
months | 4.0 [3.3 to 5.6] | 7.4 [5.7 to 7.8] | 5.6 [4.8 to 6.5]

4. Primary Outcome: Overall Survival (OS) (Phase III)
Description: OS will be evaluated by Kaplan Meier methods. The median survival and confidence intervals will be reported.
Time Frame: From study enrollment to the date of death regardless of the cause, assessed up to 5 years
Population: Eligible patients enrolled in Phase I, II and III.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 115 | 160 | 160
months | 14.5 [10.7 to 18.7] | 14.9 [12.7 to 17.1] | 12.3 [11.4 to 15.2]

5. Secondary Outcome: Objective Response Rate (ORR) (Partial or Complete Response) (Phase II)
Description: Will be assessed by RECIST v1.1 criteria. Will be tabulated by treatment group, and 95% confidence intervals presented using Wilson's Score Method. Treatment arms will be compared using a likelihood ratio chi-square test.
  Progression is defined by a 20% increase in the sum of the longest diameter of target lesions and a 5 mm absolute increase from nadir, or an unequivocal increase in a non-target lesion, or appearance of new lesions.
  For the definition of response: the responses are assessed as overall best response during the course of therapy. For partial response (PR), the sum of the longest diameters must decrease by at least 30%. For a complete response (CR), all evidence of disease must be gone and the CA125 levels must normalize. If a patient experiences a disease progression during treatment, this is classified as progressive disease (PD). If the patient neither progresses (PD) nor has a response (CR or PR), then the patient is classified as stable disease (SD).
Time Frame: Up to 5 years
Population: Eligible patients enrolled in Phase I and II.
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (PLD, Atezolizumab): A phase 3 interim futility and efficacy analysis was performed in December of 2020. This analysis recommended stopping Arm 1 (PLD+Atezo) for reasons related to futility. The public and patients were informed of the result at appropriate times. It is expected that many patients went onto non-protocol therapies in an effort to treat their condition. Any inference related to treatment efficacy or toxicity would be unreliable after this analysis.
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 88 | 88 | 88
Participants | 14 | 30 | 21

6. Secondary Outcome: ORR (Partial or Complete Response) (Phase III)
Description: Will be assessed by RECIST v1.1. Will be tabulated by treatment group, and 95% confidence intervals will be presented using Wilson's Score Method. Treatment arms will be compared using a likelihood ratio chi-square test.
  Progression is defined by a 20% increase in the sum of the longest diameter of target lesions and a 5 mm absolute increase from nadir, or an unequivocal increase in a non-target lesion, or the appearance of new lesions.
  For the definition of response: the responses are assessed as overall best response during the course of therapy. For partial response (PR), the sum of the longest diameters must decrease by at least 30%. For a complete response (CR), all evidence of disease must be gone and the CA125 levels must normalize. If a patient experiences a disease progression during treatment, this is classified as progressive disease (PD). If the patient neither progresses (PD) nor has a response (CR or PR), then the patient is classified as stable disease (SD).
Time Frame: Up to 5 years
Population: Eligible patients enrolled in Phase I, II and III.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 115 | 160 | 160
Participants | 19 | 55 | 38

7. Secondary Outcome: Number of Patients With a Grade 3 (or Higher) Adverse Event (Phase II)
Description: CTCAE V5.0 was used to classify adverse events. This endpoint will tabulate the number of patients who reported at least one adverse event of a grade 3 (or higher).
Time Frame: Up to 5 years
Population: Eligible patients enrolled in safety stage 2 or phase II and received at least one treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 84 | 88 | 86
Participants | 64 | 76 | 62

8. Secondary Outcome: Number of Patients With a Grade 3 (or Higher) Adverse Event (Phase III)
Description: as for outcome 7
Time Frame: Up to 5 years
Population: Eligible patients enrolled in safety stage 2, phase II, and phase III and received at least one treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 111 | 160 | 154
Participants | 79 | 133 | 110

9. Secondary Outcome: Patient Reported Outcomes
Description: Patient reported outcomes are measured with the NFOSI-18 Disease-related physical symptoms subscale (DRS-P). The DRS-P subscale comprises 9 items with each item ranging from 0 to 4. The total score of the DRS-P subscale ranges 0 - 36 with a larger score suggesting preferred/better health states.
Time Frame: Up to 2 years
Population: Eligible patients enrolled in Phase I, II and III and provided baseline and at least one follow-up assessments.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
Number analyzed (Participants) | 87 | 146 | 141
score
  Baseline | 26.8 (5.9) | 26.1 (6.7) | 26.3 (6.7)
  8 weeks: number analyzed (Participants) | 81 | 139 | 134
  8 weeks | 25.9 (6.3) | 25.8 (6.1) | 26.0 (5.5)
  16 weeks: number analyzed (Participants) | 73 | 118 | 107
  16 weeks | 26.8 (6.2) | 26.3 (6.3) | 26.0 (5.6)
  24 weeks: number analyzed (Participants) | 61 | 101 | 94
  24 weeks | 26.8 (6.1) | 25.7 (7.0) | 26.1 (5.7)
  32 weeks: number analyzed (Participants) | 51 | 83 | 75
  32 weeks | 26.8 (6.5) | 26.5 (6.3) | 26.4 (6.2)
  40 weeks: number analyzed (Participants) | 44 | 67 | 60
  40 weeks | 27.1 (6.8) | 27.3 (5.6) | 25.5 (5.9)
  48 weeks: number analyzed (Participants) | 42 | 64 | 50
  48 weeks | 26.8 (6.1) | 26.1 (6.1) | 25.6 (6.7)
  60 weeks: number analyzed (Participants) | 36 | 53 | 41
  60 weeks | 26.9 (6.4) | 26.7 (5.8) | 26.0 (5.4)
  72 weeks: number analyzed (Participants) | 36 | 46 | 25
  72 weeks | 27.5 (4.9) | 26.9 (5.4) | 28.8 (6.0)
  84 weeks: number analyzed (Participants) | 26 | 37 | 21
  84 weeks | 26.4 (5.6) | 27.1 (6.1) | 27.4 (5.5)
  96 weeks: number analyzed (Participants) | 20 | 30 | 15
  96 weeks | 26.6 (6.0) | 26.3 (6.4) | 29.5 (4.1)
  108 weeks: number analyzed (Participants) | 16 | 28 | 16
  108 weeks | 27.3 (6.2) | 25.0 (8.0) | 28.7 (5.6)

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: The maximum grade of each adverse event (AE) by system organ class and term (CTCAE version 5.0) will be tabulated for those individuals who at least initiate study treatment. The number and percent of subjects will be tabulated by the term.
  In order to report events potentially related to treatment, the SAE/AE population is restricted to subjects receiving treatment. The all-cause mortality is related to overall survival, which is an efficacy measure, and therefore the population is ITT.
Arm/Group | Arm I (PLD, Atezolizumab) | Arm II (PLD, Bevacizumab, Atezolizumab) | Arm III (PLD, Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 104/124 | 123/160 | 134/160
Serious Adverse Events (participants affected / at risk) | 44/111 | 86/160 | 73/154
Other Adverse Events (participants affected / at risk) | 106/111 | 159/160 | 150/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (PLD, Atezolizumab) (N=111) | Arm II (PLD, Bevacizumab, Atezolizumab) (N=160) | Arm III (PLD, Bevacizumab) (N=154)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 2 | 0
Heart failure (Cardiac disorders) | 0 | 2 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 3 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 9 | 4
Ascites (Gastrointestinal disorders) | 4 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 2 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 3
Jejunal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 9 | 1
Nausea (Gastrointestinal disorders) | 5 | 8 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 2 | 1
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 13 | 18
Small intestinal perforation (Gastrointestinal disorders) | 1 | 2 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 6 | 3
Death NOS (General disorders) | 3 | 2 | 1
Disease progression (General disorders) | 2 | 0 | 1
Edema face (General disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 6 | 2
Fever (General disorders) | 2 | 6 | 2
Flu like symptoms (General disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 2 | 0
Generalized edema (General disorders) | 0 | 1 | 0
Neck edema (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Sudden death NOS (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 5 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 3 | 1
Cardiac troponin I increased (Investigations) | 0 | 1 | 0
Cardiac troponin T increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 3 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 2
Weight loss (Investigations) | 0 | 0 | 2
White blood cell decreased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 7 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 1
Movements involuntary (Nervous system disorders) | 1 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Stroke (Nervous system disorders) | 0 | 2 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 1 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 8 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 4 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 2
Urinary fistula (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 11 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 11 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 9 | 10
Thromboembolic event (Vascular disorders) | 0 | 3 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (PLD, Atezolizumab) (N=111) | Arm II (PLD, Bevacizumab, Atezolizumab) (N=160) | Arm III (PLD, Bevacizumab) (N=154)
Anemia (Blood and lymphatic system disorders) | 55 | 62 | 63
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 5 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 7 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 12 | 5
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 3
Hearing impaired (Ear and labyrinth disorders) | 2 | 2 | 3
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 4
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 11 | 14 | 2
Hypothyroidism (Endocrine disorders) | 17 | 38 | 11
Blurred vision (Eye disorders) | 6 | 13 | 9
Cataract (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 5 | 3
Eye pain (Eye disorders) | 0 | 2 | 1
Flashing lights (Eye disorders) | 1 | 0 | 1
Floaters (Eye disorders) | 0 | 2 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Periorbital edema (Eye disorders) | 0 | 1 | 2
Photophobia (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 2 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 10 | 5 | 8
Abdominal pain (Gastrointestinal disorders) | 45 | 47 | 53
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 16 | 7 | 7
Bloating (Gastrointestinal disorders) | 15 | 14 | 13
Colitis (Gastrointestinal disorders) | 2 | 3 | 3
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 37 | 51 | 47
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 29 | 50 | 33
Dry mouth (Gastrointestinal disorders) | 6 | 5 | 8
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 13 | 10
Dysphagia (Gastrointestinal disorders) | 6 | 17 | 6
Enterocolitis (Gastrointestinal disorders) | 1 | 2 | 0
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 4 | 1
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 9 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3 | 4
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11 | 15 | 10
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 3 | 5 | 2
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2 | 3
Jejunal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 32 | 80 | 61
Nausea (Gastrointestinal disorders) | 49 | 78 | 66
Obstruction gastric (Gastrointestinal disorders) | 0 | 2 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 3 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 14 | 5
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2 | 2
Rectal mucositis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 3 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 13 | 18
Small intestinal perforation (Gastrointestinal disorders) | 0 | 2 | 1
Stomach pain (Gastrointestinal disorders) | 2 | 3 | 2
Toothache (Gastrointestinal disorders) | 1 | 4 | 4
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 33 | 56 | 40
Chills (General disorders) | 10 | 7 | 7
Edema face (General disorders) | 0 | 1 | 2
Edema limbs (General disorders) | 11 | 30 | 27
Edema trunk (General disorders) | 0 | 4 | 0
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 64 | 110 | 83
Fever (General disorders) | 18 | 23 | 7
Flu like symptoms (General disorders) | 2 | 7 | 2
Gait disturbance (General disorders) | 0 | 2 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Localized edema (General disorders) | 1 | 3 | 1
Malaise (General disorders) | 1 | 2 | 1
Neck edema (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 7 | 10
Pain (General disorders) | 9 | 20 | 14
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Allergic reaction (Immune system disorders) | 3 | 1 | 1
Bladder infection (Infections and infestations) | 0 | 0 | 1
Breast infection (Infections and infestations) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 2 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 1
Conjunctivitis infective (Infections and infestations) | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0
Esophageal infection (Infections and infestations) | 0 | 0 | 1
Gum infection (Infections and infestations) | 1 | 3 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 2 | 6 | 4
Mucosal infection (Infections and infestations) | 0 | 1 | 2
Nail infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1
Papulopustular rash (Infections and infestations) | 3 | 6 | 2
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 3 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 5 | 3
Skin infection (Infections and infestations) | 1 | 10 | 3
Tooth infection (Infections and infestations) | 0 | 9 | 1
Upper respiratory infection (Infections and infestations) | 7 | 11 | 8
Urinary tract infection (Infections and infestations) | 7 | 25 | 16
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Vulval infection (Infections and infestations) | 1 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 6 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 8 | 4
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 8 | 10
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 3
Alanine aminotransferase increased (Investigations) | 9 | 19 | 6
Alkaline phosphatase increased (Investigations) | 14 | 23 | 14
Aspartate aminotransferase increased (Investigations) | 9 | 23 | 19
Blood bilirubin increased (Investigations) | 1 | 3 | 2
Cardiac troponin I increased (Investigations) | 0 | 3 | 0
Cardiac troponin T increased (Investigations) | 0 | 2 | 0
Cholesterol high (Investigations) | 0 | 5 | 1
Creatinine increased (Investigations) | 12 | 32 | 29
Ejection fraction decreased (Investigations) | 1 | 3 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 2 | 0
GGT increased (Investigations) | 0 | 3 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 1
Hemoglobin increased (Investigations) | 0 | 1 | 0
INR increased (Investigations) | 1 | 1 | 3
Lipase increased (Investigations) | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 22 | 29 | 30
Neutrophil count decreased (Investigations) | 26 | 53 | 48
Platelet count decreased (Investigations) | 6 | 34 | 22
Serum amylase increased (Investigations) | 1 | 1 | 1
Weight gain (Investigations) | 2 | 5 | 3
Weight loss (Investigations) | 7 | 27 | 30
White blood cell decreased (Investigations) | 27 | 49 | 43
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 28 | 49 | 35
Dehydration (Metabolism and nutrition disorders) | 12 | 21 | 12
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 7 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 21 | 22 | 21
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 16 | 13
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 7 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 37 | 29
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 13 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 15 | 27 | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 18 | 10
Hyponatremia (Metabolism and nutrition disorders) | 13 | 27 | 29
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 7 | 6
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 25 | 19
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 26 | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 14 | 6
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 18 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 15 | 11
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 2 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 1 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 9 | 17 | 10
Dysarthria (Nervous system disorders) | 1 | 1 | 2
Dysesthesia (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 13 | 6
Dysphasia (Nervous system disorders) | 2 | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 23 | 54 | 33
Hypersomnia (Nervous system disorders) | 0 | 0 | 2
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 5 | 4
Movements involuntary (Nervous system disorders) | 1 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 2 | 1
Paresthesia (Nervous system disorders) | 3 | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 7 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 37 | 19
Presyncope (Nervous system disorders) | 1 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 3 | 2
Syncope (Nervous system disorders) | 1 | 3 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 2 | 3
Agitation (Psychiatric disorders) | 1 | 4 | 2
Anxiety (Psychiatric disorders) | 8 | 17 | 14
Confusion (Psychiatric disorders) | 5 | 3 | 5
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 8 | 15 | 14
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 12 | 22 | 23
Irritability (Psychiatric disorders) | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 9 | 3
Bladder spasm (Renal and urinary disorders) | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 4 | 4
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 4 | 8 | 8
Proteinuria (Renal and urinary disorders) | 7 | 36 | 31
Urinary frequency (Renal and urinary disorders) | 4 | 6 | 6
Urinary incontinence (Renal and urinary disorders) | 2 | 6 | 4
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 5 | 3
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 4 | 2
Urine discoloration (Renal and urinary disorders) | 2 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 1
Genital edema (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 4 | 4
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 4 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 4 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 4 | 4
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 2 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 39 | 31
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 | 39 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 33 | 33
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 22 | 15
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 | 13 | 9
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 9 | 6
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 12 | 11
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 5 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 28 | 85 | 51
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 23 | 9
Purpura (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 8 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 41 | 73 | 37
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 10 | 15
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 4 | 4
Flushing (Vascular disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Hot flashes (Vascular disorders) | 7 | 12 | 9
Hypertension (Vascular disorders) | 12 | 78 | 70
Hypotension (Vascular disorders) | 2 | 6 | 2
Lymphedema (Vascular disorders) | 1 | 1 | 2
Superficial thrombophlebitis (Vascular disorders) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 8 | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02839707/Prot_SAP_000.pdf